CLINICAL TRIAL: NCT02511444
Title: Intrapartum Rapid GBS Testing in Patients Presenting With Threatened Preterm Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 534-15
Record Dates: First submitted 2015-07-23; First posted 2015-07-30 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Group B Streptococcus
Keywords: GBS; GBS culture; GBS PCR; GBS colonization
MeSH Terms: interventions — Real-Time Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Other): All patients will have GBS culture and real time PCR performed.
  Interventions: Other: GBS culture and real time PCR

INTERVENTIONS:
Other: GBS culture and real time PCR — patients with signs and symptoms of threatened preterm labor, or indications for preterm delivery will have GBS colonization screened by culture and real time PCR.

SUMMARY:
The purpose of this study is to evaluate the test characteristics of a rapid intrapartum real- time polymerase chain reaction (RT-PCR) compared to the intrapartum GBS culture as the standard in preterm patients presenting with threatened preterm labor or with obstetric indications for preterm delivery.

DETAILED DESCRIPTION:
Group B streptococcus (GBS) or Streptococcus agalactiae is a gram-positive bacterium that colonizes 10-40% of maternal gastrointestinal and urogenital tract sites. Maternal colonization remains the primary risk factor and the leading cause of early onset GBS disease in infants in the United States. Transmission of GBS to the neonate in early onset GBS cases occurs at the time of labor and delivery, with a transmission rate of 52.5% if no intrapartum antibiotics are used. Of those neonates, 1-2% term infants and 8% of preterm infants will develop early onset disease.

The Centers for Disease Control (CDC) recommends universal screening at 35-37 weeks via culture of the vagina and rectum. If this is performed ≤5 weeks before delivery, it has a sensitivity of 85% and a negative predictive value of 95-98%. There is a downside to screening remote from delivery however; vaginal GBS colonization fluctuates in the same woman over time, thus rendering possibly inaccurate GBS results. It has been reported that at least 10% of antenatal GBS negative women turned positive at the time of labor. This may suggest that screening at the time of delivery is a more accurate method of predicting actual GBS colonization status. In fact, a majority of neonatal GBS sepsis occurs in infants born to mothers with a negative antepartum screening culture.

Currently, a standard GBS culture may take up to 3 days to obtain results. A rapid diagnostic test has more recently been studied as a possible method of GBS screening - real-time polymerase chain reaction (RT-PCR). Prior studies of RT-PCR, specifically the Cepheid GeneXpert GBS assay used at Miller's Children's and Women's Hospital, have reported sensitivity from 85-98.5% and specificity of 96-99.6% using data from term gestations. The CDC currently permits the use of RT-PCR as a rapid screening test for those with unknown status at term.

Several reports demonstrate that RT-PCR is a rapid, more sensitive method than standard culture for determining the intrapartum GBS colonization status. Some studies have also demonstrated the ability of RT-PCR to identify patients who would otherwise be missed by traditional GBS culture. A study by Mueller et al demonstrated that out of 64 patients with positive RT-PCR results, 10 were actually negative on culture. A cost-effectiveness analysis has demonstrated that PCR intrapartum screening strategy is not any less cost-effective than traditional culture and confers a significant decrease in early onset GBS disease in term gestations.

Preterm infants suffer the highest rate of mortality from GBS infection, with up to 30% mortality in those < 33 weeks affected by GBS sepsis. Identifying GBS colonization is thus imperative in the 7-11% of all pregnancies affected by preterm labor, given that they will not have undergone universal screening yet (which typically occurs at 35-37 weeks). While the CDC recommends giving antibiotics to patients with unknown GBS status at substantial risk for preterm delivery, implementation of this recommendation is poor.

Advantages of the RT-PCR are that its results will come back much more rapidly than the standard culture and may assist in management of these critical patients, 75 min vs 3 days, respectively. Accurate screening for GBS in a rapid fashion, especially in preterm infants, where the risk of GBS infection is most serious, can potentially allow antibiotics to be used appropriately.

The investigators seek to evaluate the utility of RT-PCR for screening of GBS in women at risk of preterm labor with an unknown GBS status. The investigators also aim to identify the ability of RT-PCR to identify GBS colonization in patients who would have otherwise been missed by culture.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Pregnant women presenting for unplanned obstetrical care at a participating clinical study site
* Gestational age between 21 6/7 and 36 6/7 weeks
* Subject has not participated in the study before
* Subject agrees to complete all aspects of the study and provide informed consent in accordance with applicable regulations
* Signs and/or symptoms suggestive of preterm labor, whereby the managing clinician suspects preterm labor
* Uterine contractions (with or without pain)
* Intermittent lower abdominal pain, dull backache, pelvic pressure
* Vaginal bleeding during the second and third trimester
* Menstrual-like intestinal cramping (with or without diarrhea)
* Change in vaginal discharge (amount, color, or consistency)
* Vague sense of discomfort characterized as "not feeling right"
* Change in cervical exam (cervical dilation, effacement, or consistency)
* Signs and symptoms necessitating preterm delivery (i.e abruption, preeclampsia, hemolysis elevated liver enzymes, low platelet (HELLP) syndrome, ruptured membranes, chorioamnionitis, fetal indications)

Exclusion Criteria:

* Exposure to antibiotics within 1 week prior to enrollment (15)
* Known GBS bacteriuria at the time of enrollment
* Prior history of neonatal GBS sepsis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2015-07; Primary Completion 2018-06 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity of intrapartum GBS real time PCR compared to intrapartum GBS culture | up to one and a half year
Positive predictive value of GBS Real time PCR performed intrapartum | up to one and a half year
Negative predictive value of GBS real time PCR performed intrapartum | up to one and a half year
Specificity of intrapartum GBS real time PCR compared to intrapartum GBS | up to one and a half year

SECONDARY OUTCOMES:
Neonatal GBS septicemia | up to one and a half year
Composite neonatal morbidity | up to one and a half year
number of neonatal intensive care unit days | up to one and a half year
Neonatal mortality rate | up to one and a half year
necrotizing enterocolitis | up to one and a half year
Gestational age at delivery | up to one and a half year
vaginal delivery | up to one and a half year
Postpartum hemorrhage | up to one and a half year
Maternal intrapartum chorioamnionitis | up to one and a half year
Maternal postpartum endometritis | up to one and a half year
Neonatal respiratory distress | up to one and half year

OTHER OUTCOMES:
Neonatal intraventricular hemorrhage | up to one and half year
Neonatal pneumonia | up to one and half year
Neonatal osteomyelitis | up to one and half year
Neonatal bacteremia | up to one and half year
Neonatal meningitis | up to one and half year
cesarean delivery | up to one and half year
composite maternal morbidity | up to one and half year

CONTACTS AND LOCATIONS:
Overall Officials: Alex Fong, MD, Principal Investigator — Maternal Fetal Medicine
Locations (1):
- Miller Children's & Women's Hospital Long Beach, Long Beach, California, United States

REFERENCES:
- [Background] Verani JR, McGee L, Schrag SJ; Division of Bacterial Diseases, National Center for Immunization and Respiratory Diseases, Centers for Disease Control and Prevention (CDC). Prevention of perinatal group B streptococcal disease--revised guidelines from CDC, 2010. MMWR Recomm Rep. 2010 Nov 19;59(RR-10):1-36. PMID 21088663
- [Background] Phares CR, Lynfield R, Farley MM, Mohle-Boetani J, Harrison LH, Petit S, Craig AS, Schaffner W, Zansky SM, Gershman K, Stefonek KR, Albanese BA, Zell ER, Schuchat A, Schrag SJ; Active Bacterial Core surveillance/Emerging Infections Program Network. Epidemiology of invasive group B streptococcal disease in the United States, 1999-2005. JAMA. 2008 May 7;299(17):2056-65. doi: 10.1001/jama.299.17.2056. PMID 18460666
- [Background] Dillon HC Jr, Gray E, Pass MA, Gray BM. Anorectal and vaginal carriage of group B streptococci during pregnancy. J Infect Dis. 1982 Jun;145(6):794-9. doi: 10.1093/infdis/145.6.794. PMID 7045248
- [Background] Regan JA, Klebanoff MA, Nugent RP. The epidemiology of group B streptococcal colonization in pregnancy. Vaginal Infections and Prematurity Study Group. Obstet Gynecol. 1991 Apr;77(4):604-10. PMID 2002986
- [Background] Turrentine MA, Ramirez MM. Recurrence of group B streptococci colonization in subsequent pregnancy. Obstet Gynecol. 2008 Aug;112(2 Pt 1):259-64. doi: 10.1097/AOG.0b013e31817f5cb9. PMID 18669720
- [Background] Hickman ME, Rench MA, Ferrieri P, Baker CJ. Changing epidemiology of group B streptococcal colonization. Pediatrics. 1999 Aug;104(2 Pt 1):203-9. doi: 10.1542/peds.104.2.203. PMID 10428995
- [Background] Valkenburg-van den Berg AW, Sprij AJ, Oostvogel PM, Mutsaers JA, Renes WB, Rosendaal FR, Joep Dorr P. Prevalence of colonisation with group B Streptococci in pregnant women of a multi-ethnic population in The Netherlands. Eur J Obstet Gynecol Reprod Biol. 2006 Feb 1;124(2):178-83. doi: 10.1016/j.ejogrb.2005.06.007. Epub 2005 Jul 18. PMID 16026920
- [Background] Gavino M, Wang E. A comparison of a new rapid real-time polymerase chain reaction system to traditional culture in determining group B streptococcus colonization. Am J Obstet Gynecol. 2007 Oct;197(4):388.e1-4. doi: 10.1016/j.ajog.2007.06.016. PMID 17904971
- [Background] Puopolo KM, Madoff LC, Eichenwald EC. Early-onset group B streptococcal disease in the era of maternal screening. Pediatrics. 2005 May;115(5):1240-6. doi: 10.1542/peds.2004-2275. PMID 15867030
- [Background] Young BC, Dodge LE, Gupta M, Rhee JS, Hacker MR. Evaluation of a rapid, real-time intrapartum group B streptococcus assay. Am J Obstet Gynecol. 2011 Oct;205(4):372.e1-6. doi: 10.1016/j.ajog.2011.06.087. Epub 2011 Jun 29. PMID 21864820
- [Background] Goins WP, Talbot TR, Schaffner W, Edwards KM, Craig AS, Schrag SJ, Van Dyke MK, Griffin MR. Adherence to perinatal group B streptococcal prevention guidelines. Obstet Gynecol. 2010 Jun;115(6):1217-1224. doi: 10.1097/AOG.0b013e3181dd916f. PMID 20502293
- [Background] Van Dyke MK, Phares CR, Lynfield R, Thomas AR, Arnold KE, Craig AS, Mohle-Boetani J, Gershman K, Schaffner W, Petit S, Zansky SM, Morin CA, Spina NL, Wymore K, Harrison LH, Shutt KA, Bareta J, Bulens SN, Zell ER, Schuchat A, Schrag SJ. Evaluation of universal antenatal screening for group B streptococcus. N Engl J Med. 2009 Jun 18;360(25):2626-36. doi: 10.1056/NEJMoa0806820. PMID 19535801
- [Background] de Tejada BM, Pfister RE, Renzi G, Francois P, Irion O, Boulvain M, Schrenzel J. Intrapartum Group B streptococcus detection by rapid polymerase chain reaction assay for the prevention of neonatal sepsis. Clin Microbiol Infect. 2011 Dec;17(12):1786-91. doi: 10.1111/j.1469-0691.2010.03378.x. Epub 2011 Apr 12. PMID 20860701
- [Background] Edwards RK, Novak-Weekley SM, Koty PP, Davis T, Leeds LJ, Jordan JA. Rapid group B streptococci screening using a real-time polymerase chain reaction assay. Obstet Gynecol. 2008 Jun;111(6):1335-41. doi: 10.1097/AOG.0b013e31817710ee. PMID 18515517
- [Background] El Helali N, Nguyen JC, Ly A, Giovangrandi Y, Trinquart L. Diagnostic accuracy of a rapid real-time polymerase chain reaction assay for universal intrapartum group B streptococcus screening. Clin Infect Dis. 2009 Aug 1;49(3):417-23. doi: 10.1086/600303. PMID 19580414
- [Background] Convert M, Martinetti Lucchini G, Dolina M, Piffaretti JC. Comparison of LightCycler PCR and culture for detection of group B streptococci from vaginal swabs. Clin Microbiol Infect. 2005 Dec;11(12):1022-6. doi: 10.1111/j.1469-0691.2005.01275.x. PMID 16307558
- [Background] Davies HD, Miller MA, Faro S, Gregson D, Kehl SC, Jordan JA. Multicenter study of a rapid molecular-based assay for the diagnosis of group B Streptococcus colonization in pregnant women. Clin Infect Dis. 2004 Oct 15;39(8):1129-35. doi: 10.1086/424518. Epub 2004 Sep 14. PMID 15486835
- [Background] Goodrich JS, Miller MB. Comparison of culture and 2 real-time polymerase chain reaction assays to detect group B Streptococcus during antepartum screening. Diagn Microbiol Infect Dis. 2007 Sep;59(1):17-22. doi: 10.1016/j.diagmicrobio.2007.03.023. Epub 2007 May 16. PMID 17509794
- [Background] Rallu F, Barriga P, Scrivo C, Martel-Laferriere V, Laferriere C. Sensitivities of antigen detection and PCR assays greatly increased compared to that of the standard culture method for screening for group B streptococcus carriage in pregnant women. J Clin Microbiol. 2006 Mar;44(3):725-8. doi: 10.1128/JCM.44.3.725-728.2006. PMID 16517846
- [Background] Mueller M, Henle A, Droz S, Kind AB, Rohner S, Baumann M, Surbek D. Intrapartum detection of Group B streptococci colonization by rapid PCR-test on labor ward. Eur J Obstet Gynecol Reprod Biol. 2014 May;176:137-41. doi: 10.1016/j.ejogrb.2014.02.039. Epub 2014 Mar 12. PMID 24680393
- [Background] El Helali N, Giovangrandi Y, Guyot K, Chevet K, Gutmann L, Durand-Zaleski I. Cost and effectiveness of intrapartum group B streptococcus polymerase chain reaction screening for term deliveries. Obstet Gynecol. 2012 Apr;119(4):822-9. doi: 10.1097/AOG.0b013e31824b1461. PMID 22433346
- [Background] Wernecke M, Mullen C, Sharma V, Morrison J, Barry T, Maher M, Smith T. Evaluation of a novel real-time PCR test based on the ssrA gene for the identification of group B streptococci in vaginal swabs. BMC Infect Dis. 2009 Sep 4;9:148. doi: 10.1186/1471-2334-9-148. PMID 19732424